CLINICAL TRIAL: NCT04204343
Title: Comparing Analgesic Effects of Ultrasound-Guided Caudal and Erector Spinae Plane Blocks in Pediatric Patients Undergoing Upper Abdominal Surgery: A Randomized Controlled Double-Blinded Study
Brief Title: Comparing Analgesic Effects of Caudal and Erector Spinae Plane Blocks in Pediatrics Undergoing Upper Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2018/1073
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Anesthesia, Local
Keywords: Erector Spinae Plane Block; Caudal Block; Ultrasound guidance; Postoperative analgesia; Upper abdominal surgery
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: RANDOMISED DOUBLE BLINDED INTERVENTIONAL
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal Block (Active Comparator): US-guided caudal block with 0.7 ml/kg 0.25% Bupivacaine
  Interventions: Drug: Bupivacaine 0.7 ml/kg
- Erector Spinae Plane Block (Active Comparator): US-guided erector spinae plane block with 0.5 ml/kg 0.25% Bupivacaine
  Interventions: Drug: Bupivacaine 0.5 ml/kg

INTERVENTIONS:
Drug: Bupivacaine 0.7 ml/kg — Bupivacaine 0.25% 0.7 ml/kg
  Other Names: Marcaine
  Arms: Caudal Block
Drug: Bupivacaine 0.5 ml/kg — Bupivacaine 0.25% 0.5 ml/kg
  Other Names: Marcaine
  Arms: Erector Spinae Plane Block

SUMMARY:
Upper abdominal surgeries are painful and pediatric patients who undergo these operations require effective postoperative pain control. Epidural and caudal blocks are considered to be the gold standard regional analgesia techniques. Currently, ultrasound guidance is commonly used for caudal block performances to demonstrate the cannula placement and the deposition of local anesthetic. Additionally, erector spinae plane block can be a safer alternative for blocking the similar dermatomes. In this study, the aim is to compare postoperative analgesic effects of these two ultrasound-guided techniques in pediatric patients. The primary outcome of this study is the follow-up of FLACC/VAS pain scores. Secondary outcomes are time to first analgesic requirement, number of patients who require rescue analgesic, possible side effects, time to first mobilization, length of hospital stay and chronic pain due to incision after 2 months.

DETAILED DESCRIPTION:
Upper abdominal surgeries are painful and pediatric patients who undergo these operations require effective postoperative pain control. Blockade of dermatomes between T6 and L1 commonly provides effective postoperative analgesia. Epidural and caudal blocks are considered to be the gold standard regional analgesia techniques as they provide both somatic and visceral analgesia. Currently, ultrasound guidance is commonly used for caudal block performances to demonstrate the cannula placement and the deposition of local anesthetic. Additionally, erector spinae plane block can be a safer alternative for blocking the similar dermatomes. In the present study, the aim is to compare postoperative analgesic effects of these two ultrasound-guided techniques in pediatric patients undergoing upper abdominal surgery. The primary outcome of this study is the follow-up of FLACC/VAS pain scores. Secondary outcomes are time to first analgesic requirement, number of patients who require rescue analgesic, possible side effects (nausea, vomiting, itching, urinary retention, bradycardia, hypotension, respiratory depression), time to first mobilization, length of hospital stay and chronic pain due to incision after 2 months.

ELIGIBILITY:
Inclusion Criteria:

* undergoing upper abdominal surgery
* ASA(American Society of Anesthesiology)1-2

Exclusion Criteria:

* denial of patient or parents
* infection on the local anesthetic application area
* infection in the central nervous system
* coagulopathy
* brain tumors
* known allergy against local anesthetics
* anatomical difficulties
* with preexisting cardiac dysfunction
* with history of renal and/or hepatic dysfunction

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
The Face, Legs, Activity, Cry, Consolability scale/Visual Analog scale | up to 48 hours
  Pain scores between 0-10

SECONDARY OUTCOMES:
length of hospital stay | through study completion, an average of 1 week
  hospitalisation
number patients who require rescue analgesic | up to 48 hours
  number of patients who require IV morphine (0.03 mg/kg) during the first 2 hours and paracetamol in the 48 hours
Time to first analgesic | up to 48 hours
  Duration of postoperative analgesia
Incidence of side effects/complications | up to first week
  hematoma, dural puncture, infections
Time to first mobilization | up to 48 hours
  time to first mobilization
Presence of pain (chronic pain - Visual Analog scale>3) | 3 months
  Chronic pain due to incision after 2-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, Principal Investigator — Istanbul University Faculty of Medicine Department of Anesthesiology
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Ultrasound-Guided Single-Shot Preemptive Erector Spinae Plane Block for Postoperative Pain Management. — https://www.ncbi.nlm.nih.gov/pubmed/30477888
- See also: Erector Spinae Plane Block in Management of Pain After Kidney Transplantation. — https://www.ncbi.nlm.nih.gov/pubmed/30412258
- See also: The Erector Spinae Plane Block. — https://www.ncbi.nlm.nih.gov/pubmed/28207652
- See also: Caudal Epidural Block: An Updated Review of Anatomy and Techniques. — https://www.ncbi.nlm.nih.gov/pubmed/28337460
- See also: Expert opinion: regional nerve blocks in everyday pediatric urology: 2. Ultrasound-guided regional anesthetic caudal block. — https://www.ncbi.nlm.nih.gov/pubmed/30502063